CLINICAL TRIAL: NCT05279729
Title: Efficacy of mHealth Apps for Health in a Low-income, Type II Diabetic, Hispanic
Brief Title: Efficacy of mHealth Apps for Health in a Low-income, Type II Diabetic, Hispanic Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HS-2021-0245
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: diabetes; low income; mhealth; ehealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Weight Watchers (WW) (Experimental)
  Interventions: Other: Mobile health application
- Healthi app (Experimental)
  Interventions: Other: Mobile health application

INTERVENTIONS:
Other: Mobile health application — Intervention will be with two different mobile health (mHealth) applications, Weight Watchers and Healthi app (formerly iTrackBites)
  Arms: Healthi app; Weight Watchers (WW)

SUMMARY:
The purpose of this study is to determine the effectiveness of mobile health applications in improving health outcomes and the subsequent benefit of improving type II diabetes outcomes in a low socioeconomic Hispanic population. This study will involve a 6-month long commitment where participants will be expected to weigh themselves every morning, at the same time, and check their blood glucose readings daily before and after meals for at least three meals in the day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type II diabetes
* Between the age of 18-64
* BMI ≥ 27
* Individual annual income less than $47,520 [Covered CA income guidelines and salary restrictions]
* Hispanic and/or Latinx origin
* Monitors blood glucose regularly
* Owns or has access to a bathroom weight scale
* Owns a smartphone and willing to download mobile apps

Exclusion Criteria:

* Does not check blood glucose at least once per day
* On medications that promote weight gain such as antipsychotic, antidepressant, and steroid hormone medications.

Medications for diabetes such as insulin, thiazolidinediones or sulfonylureas are okay

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of mHealth apps at reducing bodyweight assessed by bodyweight measurements over 6 months | 6 months
  Determine if mHealth apps-Weight Watchers (WW) and Healthi app-are an effective weight loss modality compared to standard weight loss program (control)
Most effect intervention for weight loss in first 3 months | 6 months
  Compare the three interventions, mHealth apps and control, against each other to determine which is most effective at achieving the maximum amount of weight loss within the first three months
Most effective intervention for weight loss by 6 months | 6 months
  Compare and determine which intervention leads to the highest weight loss maintenance after six months
Self-efficacy in weight management assessed by Weight Management and Nutrition Knowledge questionnaire | 6 months
  Compare and determine which intervention promotes self-efficacy in weight management
Long term diabetes improvement via A1c | 6 months
  Compare and determine which intervention provides the best improvements towards diabetes via blood glucose and HbA1c

SECONDARY OUTCOMES:
Quality of Life after using mHealth apps assessed by World Health Organization Quality of Life BREF questionnaire | 6 months
  Comparing the three interventions to determine which leads to greater quality of life (QOL)
mhealthy app preference assessed by questionnaire | 6 months
  Which mHealth app is more economically feasible for the participants and if feasibility changes after app usage. Outcome will be assessed with a questionnaire asking if the participant can afford the app.

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No